CLINICAL TRIAL: NCT02280382
Title: An Intervention to Improve the Management of Posterior Vaginal Compartment Prolapse Using Femmeze®: a Feasibility Study
Brief Title: An Intervention to Improve Prolapse Using Femmeze® (v1)
Acronym: Femmeze®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Cornwall Hospitals Trust (Other)
Collaborators: Peninsula Health (Other Government)
Responsible Party: Principal Investigator, Sharon Eustice, Nurse Consultant, Royal Cornwall Hospitals Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014.RCHT.76
Record Dates: First submitted 2014-10-15; First posted 2014-10-31 (Estimated); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Rectocele; Pelvic Organ Prolapse
Keywords: splinting
MeSH Terms: conditions — Rectocele; Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Femmeze® (Other): Femmeze® will be used by women in the intervention group for 8 weeks These women will be measuring against their usual care in a linear design; measurement will include validated questionnaires
  Interventions: Device: Femmeze®

INTERVENTIONS:
Device: Femmeze® — Femmeze will be used by women in the intervention group for 8 weeks These women will be measuring against their usual care in a linear design; measurement will include validated questionnaires
  Other Names: 5060228630194

SUMMARY:
The main purpose of the feasibility study is to identify the patient experience of Femmeze® which is a device aimed at improving posterior vaginal compartment prolapse (rectocele) for women with obstructive defaecation. The investigators want to investigate implementation and preliminary effectiveness of the device. The method of investigation will be a pre-post intervention design, which involves asking 30 women to use Femmeze® over a period of 8 weeks. This is an academic study on a labelled indication (http://www.nres.nhs.uk/search/?q=medical+devices).

DETAILED DESCRIPTION:
Aim Evaluate the feasibility of the Femmeze® device to improve management of posterior vaginal compartment prolapse addressing implementation of the intervention and preliminary effectiveness.

Objectives

* demonstrate effectiveness of the device (comfort, ease of use, empty the rectum of stool more easily than their current approach and quality of life)
* identify which stage of prolapse the device would be most suitable
* identify any changes to the device or instructions for use (needs adjustment to its design in terms of length/width)

The study will use a pre-post intervention design with the aim of evaluating the feasibility of the intervention (using the device); and identifying any implementation issues and preliminary effectiveness. The participants will be followed prospectively to compare the device against their own usual care. Usual care in this context will be using their fingers to help empty their rectum of stool.

Participants will be invited to complete a semi-structured interview to understand their lived experience. A Patient and Public Involvement Group has contributed to improving the study methods.

ELIGIBILITY:
Inclusion Criteria:

* Adult women (over 18 years of age) with symptoms of obstructive defaecation
* Not undergone posterior vaginal compartment prolapse surgery

Exclusion Criteria:

* Cognitive impairment
* Hand disability
* Refuse to give informed consent
* Pregnancy
* Less than 12 weeks post-partum
* Neurological disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Quality of life instrument (ICIQ-Vaginal Symptoms) | 12 months
  http://www.iciq.net/ICIQ-VS.html

SECONDARY OUTCOMES:
Device feedback questionnaire | 12 months
  evaluating the device from the participants perspective

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Eustice, BSc; MSc, Principal Investigator — RCHT
Locations (1):
- RoyalCornwallHT, Truro, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes